CLINICAL TRIAL: NCT06931561
Title: Occupational Cancer Screening in Firefighters: A Pilot Study Within the Inova Health System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Collaborators: Virginia Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: INOVA-2024-320
Record Dates: First submitted 2025-03-28; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Whole Body MRI (Active Comparator): Prenuvo whole body magnetic resonance imaging
  Interventions: Procedure: Whole Body MRI; Device: MCD Assay; Other: Occupational Exposure Questionnaire
- Whole Body Ultrasound (Active Comparator): High frequency sound waves
  Interventions: Procedure: Whole Body Ultrasound; Device: MCD Assay; Other: Occupational Exposure Questionnaire

INTERVENTIONS:
Procedure: Whole Body MRI — Whole body MRI
  Arms: Whole Body MRI
Procedure: Whole Body Ultrasound — Whole Body Ultrasound
  Arms: Whole Body Ultrasound
Device: MCD Assay — Cancer detection blood test
Other: Occupational Exposure Questionnaire — Questionnaire

SUMMARY:
The purpose of this study is to further understand the clinical impact and follow-up steps that may be required based on using whole-body Magnetic Resonance Imaging (MRI) or whole-body ultrasound and blood tests to detect multiple cancers in firefighters.

This study involves an investigational test (cancer blood test) that has not been approved by the U.S. Food and Drug Administration (FDA).

Whole-body MRI and whole-body ultrasound are approved by the U.S. Food and Drug Administration (FDA) to be used in the diagnosis of some cancers and is approved for adults and children who present other signs of potential disease. In this study, however, the whole-body MRI and the whole-body ultrasound are considered investigational devices because they are not yet approved for use in healthy adults with no other cancer indications.

DETAILED DESCRIPTION:
In July 2022, a Working Group of the International Agency for Research on Cancer (IARC) concluded that occupational work as a firefighter is carcinogenic to humans (Group 1) based on a comprehensive review of the scientific literature. Given the established higher risk of multiple cancer types in firefighters, an emphasis on evaluating and delivering evidence-based preventive health services including screening for early detection of cancer in this population is imperative. Evidence-based recommendations on the optimal screening approach for firefighters at higher risk of cancer and greater understanding of the risks and benefits of investigational screening modalities that firefighters are currently receiving in real-world practice are needed. As part of a multidisciplinary cancer screening program for firefighters that is being conducted by the Saville Cancer Screening and Prevention Center and Department of Occupational Health within the Inova Health System, the purpose of this research study is to generate preliminary data on the clinical impact of investigational cancer screening modalities in 800 career and volunteer firefighters age ≥ 35 years old with at least 10 cumulative years of employment as a firefighter. Participating firefighters will be randomized equally to one of two whole-body imaging screening arms (1. whole body MRI, 2. whole body ultrasound) and all participants will further be screened with a multi-cancer detection assay. Aims include evaluating the clinical impact and performance of each tool in detecting cancer, the diagnostic follow-up and healthcare utilization prompted by use of each investigational tool, and assessments of anxiety and feasibility of implementation related to the screening protocols in participants. It is anticipated that results from this pilot will support the development of future firefighter cancer screening programs and serve as a research framework that can be adopted and tested within other health systems in partnership with the local fire jurisdictions in their catchment area, with the ultimate goal of identifying the risks and benefits of these tools for early cancer detection in the firefighter population.

All whole-body MRI examinations will be conducted without contrast using 1.5T (T is a unit of measure for magnetic field strength) (Tesla) MRI systems (Philips Healthcare Clinical Systems, Amsterdam, Netherlands). Scans will be obtained at an outpatient MRI facility with the images subsequently reviewed and reported by the imaging center radiologists specialized in the practice of preventive healthcare screening using whole-body MRI. The scan protocol that will be used for this research study is designed to be consistent with the protocol that has been implemented at external imaging centers such as Prenuvo where firefighters are already being screened. The resulting whole-body MRI report and images will be sent to the Saville clinical team who will use the report from the consulting radiologist to determine the follow-up diagnostic plan, as appropriate. The imaging report will include an interpretation of findings from each organ system with an assessment based on the Oncologically Relevant Findings Reporting and Data System (ONCO-RADS) along with any applicable clinical notes from the reviewing radiologist.

Whole-Body Ultrasound:

All whole-body ultrasound examinations will be conducted by a vendor that specializes in ultrasound diagnostics using the Mindray Z60 ultrasound technology with site-specific presets. The procedure will include scans of the liver, spleen, gallbladder, kidneys, thyroid (scanning of the right and left lobes of the gland to evaluate any nodules or echotexture changes), heart, and bladder. For female patients, further evaluation of the reproductive system including the uterus and ovaries will be assessed transabdominally while the urinary bladder is at its fullest capacity. For male patients, imaging of the testicles and surrounding region will also be performed. Any abnormality detected during the scan will be imaged multiple times with and without color (color imaging is used to show vascularity in the region where an abnormality is noted). Identical protocols and procedures for this scan will be used for all participants randomized to receive wholebody ultrasound and will be performed by the same imaging company. Unified Diagnostic Services (UDS), the ultrasound vendor, will provide the mobile ultrasounds at a location convenient to the participants, which could include the Saville Cancer Screening and Prevention Center, an Inova Occupational Health location, or directly at the firehouse or other convenient community location of a participating jurisdiction.

Multiple Cancer Detection (MCD) Test:

Blood samples collected from all participants for this assay (Cancerguard EXTM) will be shipped to and analyzed at the central laboratory of the collaborating MCD company. Blood draws will be collected either at the Saville Cancer Screening and Prevention Center by clinical research staff, or using mobile phlebotomy at a location outside of the Saville Center that is convenient for the firefighter (e.g., Inova Occupational Health location, firehouse at the participating jurisdiction). The assay may include whole or targeted genetic sequencing to sequence healthy DNA or abnormal DNA. A study report indicating whether a cancer signal has been detected from analysis of the blood sample will be issued to the Saville Center clinical investigators. For participants that do not have a cancer signal detected, no further diagnostic evaluations will be scheduled based on this particular screening test. Participants who do have a cancer signal detected will undergo diagnostic follow-up as clinically appropriate. In rare cases, there may be an invalid test results due to sample collection and/or processing errors. Participants with and invalid test results will have the option to undergo a repeat blood draw. If a participant declines the repeat blood draw, the invalid test result will not terminate the participant from the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 35 years old
* at least 10 cumulative years working as a firefighter
* Completion of National Fire Protection Association (NFPA) physical examination within the past 6 months for active-duty firefighters (retired firefighters do not need to meet this criteria)
* Ability to understand and willing to sign informed consent
* Ability to understand and willing to sign the Health Insurance Portability and Accountability Act (HIPAA) Authorization
* Additional eligibility criteria in protocol

Exclusion Criteria:

* No prior history of any invasive cancer within the previous 5 years (non-melanoma skin cancer and in situ carcinoma would still be eligible) and no current diagnostic workup for suspicion of cancer.
* Received a whole-body MRI, whole-body ultrasound, or been tested with a MCD within the past 1-year
* For women of childbearing potential, pregnancy
* Additional exclusion criteria in protocol

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of confirmed pre-malignancies detected with each investigational screening tool | up to 1 year (± 2 months)
  The number of confirmed pre-malignancies detected using whole-body Magnetic Resonance Imaging (MRI), whole-body ultrasound, or the Multi Cancer Detection (MCD) test
Number of confirmed malignancies detected with each investigational screening tool | up to 1 year (± 2 months)
  The number of confirmed malignancies detected using whole-body Magnetic Resonance Imaging (MRI), whole-body ultrasound, or the Multi Cancer Detection (MCD) test

OTHER OUTCOMES:
Sensitivity of each investigational screening tool | up to 1 year (± 2 months)
  Sensitivity of each investigational screening tool (whole-body ultrasound, whole-body MRI, and MCD test)
Specificity of each investigational screening tool | up to 1 year (± 2 months)
  Specificity of each investigational screening tool (whole-body ultrasound, whole-body MRI, and MCD test)
Negative predictive value (NPV) of each investigational screening tool | up to 1 year (± 2 months)
  Negative predictive value (NPV) of each investigational screening tool (whole-body ultrasound, whole-body MRI, and MCD test)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Van Bebber, Study Director — Inova Health System - Inova Schar Cancer; Rebecca Kaltman, MD, Principal Investigator — Inova Health System - Saville Cancer Screening and Prevention Center
Locations (1):
- Inova Schar Cancer - Saville Cancer Screening and Prevention Center, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
All data and records generated during this study will be kept confidential in accordance with Inova Health System institutional policies and HIPAA on participant privacy. The Investigator and other site personnel will not use such data and records for any purpose other than conducting the study. No identifiable data will be shared with anyone outside of the authorized Investigators and clinical research staff involved in the study. It is possible that aggregate data results from the project may be shared with other researchers in the future to facilitate pooled analyses or meta-analyses. Individual patient-level data will not be shared.

REFERENCES:
- [Background] LeMasters GK, Genaidy AM, Succop P, Deddens J, Sobeih T, Barriera-Viruet H, Dunning K, Lockey J. Cancer risk among firefighters: a review and meta-analysis of 32 studies. J Occup Environ Med. 2006 Nov;48(11):1189-202. doi: 10.1097/01.jom.0000246229.68697.90. PMID 17099456
- [Background] Jalilian H, Ziaei M, Weiderpass E, Rueegg CS, Khosravi Y, Kjaerheim K. Cancer incidence and mortality among firefighters. Int J Cancer. 2019 Nov 15;145(10):2639-2646. doi: 10.1002/ijc.32199. Epub 2019 Mar 1. PMID 30737784
- [Background] Demers PA, DeMarini DM, Fent KW, Glass DC, Hansen J, Adetona O, Andersen MH, Freeman LEB, Caban-Martinez AJ, Daniels RD, Driscoll TR, Goodrich JM, Graber JM, Kirkham TL, Kjaerheim K, Kriebel D, Long AS, Main LC, Oliveira M, Peters S, Teras LR, Watkins ER, Burgess JL, Stec AA, White PA, DeBono NL, Benbrahim-Tallaa L, de Conti A, El Ghissassi F, Grosse Y, Stayner LT, Suonio E, Viegas S, Wedekind R, Boucheron P, Hosseini B, Kim J, Zahed H, Mattock H, Madia F, Schubauer-Berigan MK. Carcinogenicity of occupational exposure as a firefighter. Lancet Oncol. 2022 Aug;23(8):985-986. doi: 10.1016/S1470-2045(22)00390-4. Epub 2022 Jul 1. No abstract available. PMID 35780778
- [Background] Pinkerton L, Bertke SJ, Yiin J, Dahm M, Kubale T, Hales T, Purdue M, Beaumont JJ, Daniels R. Mortality in a cohort of US firefighters from San Francisco, Chicago and Philadelphia: an update. Occup Environ Med. 2020 Feb;77(2):84-93. doi: 10.1136/oemed-2019-105962. Epub 2020 Jan 2. PMID 31896615
- [Background] Daniels RD, Bertke S, Dahm MM, Yiin JH, Kubale TL, Hales TR, Baris D, Zahm SH, Beaumont JJ, Waters KM, Pinkerton LE. Exposure-response relationships for select cancer and non-cancer health outcomes in a cohort of U.S. firefighters from San Francisco, Chicago and Philadelphia (1950-2009). Occup Environ Med. 2015 Oct;72(10):699-706. doi: 10.1136/oemed-2014-102671. Epub 2015 Feb 11. PMID 25673342
- [Background] DeBono NL, Daniels RD, Beane Freeman LE, Graber JM, Hansen J, Teras LR, Driscoll T, Kjaerheim K, Demers PA, Glass DC, Kriebel D, Kirkham TL, Wedekind R, Filho AM, Stayner L, Schubauer-Berigan MK. Firefighting and Cancer: A Meta-analysis of Cohort Studies in the Context of Cancer Hazard Identification. Saf Health Work. 2023 Jun;14(2):141-152. doi: 10.1016/j.shaw.2023.02.003. Epub 2023 Mar 7. PMID 37389311
- [Background] Kwee RM, Kwee TC. Whole-body MRI for preventive health screening: A systematic review of the literature. J Magn Reson Imaging. 2019 Nov;50(5):1489-1503. doi: 10.1002/jmri.26736. Epub 2019 Apr 1. PMID 30932247
- [Background] Kim A, Chung KC, Keir C, Patrick DL. Patient-reported outcomes associated with cancer screening: a systematic review. BMC Cancer. 2022 Mar 1;22(1):223. doi: 10.1186/s12885-022-09261-5. PMID 35232405
- [Background] Summers P, Saia G, Colombo A, Pricolo P, Zugni F, Alessi S, Marvaso G, Jereczek-Fossa BA, Bellomi M, Petralia G. Whole-body magnetic resonance imaging: technique, guidelines and key applications. Ecancermedicalscience. 2021 Jan 7;15:1164. doi: 10.3332/ecancer.2021.1164. eCollection 2021. PMID 33680078
- [Background] Zugni F, Padhani AR, Koh DM, Summers PE, Bellomi M, Petralia G. Whole-body magnetic resonance imaging (WB-MRI) for cancer screening in asymptomatic subjects of the general population: review and recommendations. Cancer Imaging. 2020 May 11;20(1):34. doi: 10.1186/s40644-020-00315-0. PMID 32393345
- [Background] Lee SY, Park HJ, Kim MS, Rho MH, Han CH. An initial experience with the use of whole body MRI for cancer screening and regular health checks. PLoS One. 2018 Nov 21;13(11):e0206681. doi: 10.1371/journal.pone.0206681. eCollection 2018. PMID 30462666
- [Background] Consul N, Amini B, Ibarra-Rovira JJ, Blair KJ, Moseley TW, Taher A, Shah KB, Elsayes KM. Li-Fraumeni Syndrome and Whole-Body MRI Screening: Screening Guidelines, Imaging Features, and Impact on Patient Management. AJR Am J Roentgenol. 2021 Jan;216(1):252-263. doi: 10.2214/AJR.20.23008. Epub 2020 Nov 5. PMID 33151095
- [Background] Hu YS, Wu CA, Lin DC, Lin PW, Lee HJ, Lin LY, Lin CJ. Applying ONCO-RADS to whole-body MRI cancer screening in a retrospective cohort of asymptomatic individuals. Cancer Imaging. 2024 Feb 7;24(1):22. doi: 10.1186/s40644-024-00665-z. PMID 38326850
- [Background] Geiger KW, Wright TJ, Deters L. Renal Cell Carcinoma as an Incidental Finding in Firefighters: A Case Series. Cureus. 2020 Jul 18;12(7):e9259. doi: 10.7759/cureus.9259. PMID 32821605
- [Background] Printz C. New research finds lung cancer screening guidelines are insufficient for firefighters. Cancer. 2020 Feb 15;126(4):692-693. doi: 10.1002/cncr.32721. No abstract available. PMID 31995245
- [Background] Rubinstein WS, Patriotis C, Dickherber A, Han PKJ, Katki HA, LeeVan E, Pinsky PF, Prorok PC, Skarlupka AL, Temkin SM, Castle PE, Minasian LM. Cancer screening with multicancer detection tests: A translational science review. CA Cancer J Clin. 2024 Jul-Aug;74(4):368-382. doi: 10.3322/caac.21833. Epub 2024 Mar 22. PMID 38517462
- [Background] Brito-Rocha T, Constancio V, Henrique R, Jeronimo C. Shifting the Cancer Screening Paradigm: The Rising Potential of Blood-Based Multi-Cancer Early Detection Tests. Cells. 2023 Mar 18;12(6):935. doi: 10.3390/cells12060935. PMID 36980276
- [Background] Petralia G, Koh DM, Attariwala R, Busch JJ, Eeles R, Karow D, Lo GG, Messiou C, Sala E, Vargas HA, Zugni F, Padhani AR. Oncologically Relevant Findings Reporting and Data System (ONCO-RADS): Guidelines for the Acquisition, Interpretation, and Reporting of Whole-Body MRI for Cancer Screening. Radiology. 2021 Jun;299(3):494-507. doi: 10.1148/radiol.2021201740. Epub 2021 Apr 27. PMID 33904776
- See also: International Agency for Research on Cancer. IARC Monographs Firefighting — https://publications.iarc.fr/615